CLINICAL TRIAL: NCT02727985
Title: Opioid Reduction Following Spinal Cord Stimulation: A Comparison of Two Protocols, Effect on Patient Quality of Life and Cost-Impact to the Healthcare System
Brief Title: Opioid Reduction Following Spinal Cord Stimulation
Acronym: REDUCE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Site did not meet recruitment goals and target numbers
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB15-118
Record Dates: First submitted 2016-03-18; First posted 2016-04-05 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist weaning schedule (Experimental): The Neuromodulation clinic pharmacist will develop a weaning schedule for these patients. Schedules will be individualized taking into account the amount of opioid, duration of opioid use, other adjunctive medications, and specific variables related to the patient.
  Interventions: Procedure: Pharmacist weaning schedule
- Self/Family Physician weaning schedule (No Intervention): Patients will wean off their opioids by themselves or with their family physician without the assistance of a prepared schedule.

INTERVENTIONS:
Procedure: Pharmacist weaning schedule — individualized weaning schedule for each patient taking into account the amount of opioid, duration of opioid use, other adjunctive medications, and specific variables related to the patient.
  Arms: Pharmacist weaning schedule

SUMMARY:
The primary purpose of this study is to compare opioid use post-spinal cord stimulation implant at 1, 3, 6, 9 and 12 month intervals in patients who were provided with a weaning schedule by the Neuromodulation team (experimental group) versus those who wean on their own or with their family doctor (control group; standard care) to determine if one strategy is superior to the other.

The secondary objectives will be to further characterize change in opioid use as it relates to pain scores, quality of life and disability from baseline to follow-up assessments. The investigators will examine changes in opioid-related adverse events and medication costs to help understand the impact of opioid weaning on the patient and the system. The investigators will also compare worker's compensation patients with non-worker compensation patients to see if they follow the same result pattern.

DETAILED DESCRIPTION:
The Neuromodulation clinic in the Regina Qu'Appelle Health Region currently provides service to 501 patients with 266 of those being spinal cord stimulation (SCS) cases. There is an average of 30 new SCS cases per year with the majority of those being implanted for unilateral or bilateral leg pain with or without low back pain. All patients are done via a two-step process consisting of an initial trial with an externalized electrode for a 1-2 week trial period. At the end of the trial period, if successful, the patient undergoes the internalization procedure. Our goal during the trial period is to achieve a pain reduction of 50% or more. Our mean success rates for trial to implant are approximately 80%. After the internalization procedure, patients are instructed to slowly begin weaning their pain medications.

There is scant data discussing the effect of SCS systems on medication use and particularly, opioids. To date, pain medication weaning has been largely left to the discretion of the patient with no formalized system for oversight. This has resulted in poor rates of reduction of opioid consumption in spite of improved pain relief achieved with SCS. In addition, should a patient have a successful SCS trial and move on to the permanent implant, how do we break them of their dependence on opioids? Some patients have a good relationship with their family physician and will rely on him/her to help wean them off the opioids. Others feel that they can manage weaning on their own (self-management). As intensity of pain improves along with quality of life, pain medication consumption should decrease in tandem without jeopardizing pain control. However, a lack of adherence by the patient or family physician would interfere with this process. The current standard of care is for the patient and their family physician to decide the best weaning process. The investigators propose that having a multidisciplinary Neuromodulation team with a dedicated pharmacist who can draw up a patient specific weaning schedule and follow the patient closely would more effectively reduce opioid consumption than patient (self-management) or family physician-aided weaning alone

Importance of this Study Chronic pain is estimated to cost the Canadian health care system $6 billion per year according to the Canadian Pain Society with this number expected to continue to rise. SCS systems have been proven to be more cost effective than conventional medical management for chronic pain patients. Increased use of SCS systems would help to decrease the burden on our health care dollars. In addition, the added risk of long term opioid use leads to issues of tolerance, physical dependence and potential adverse effects including overdose. Social concerns regarding opioid divergence and inappropriate use must also be taken into account. The goal for this project is to further strengthen the support for the use of SCS and provide information on the most effective way to decrease opioid use among the chronic pain population.

Research Purpose and Objectives:

The primary purpose of this study is to compare opioid use post-SCS implant at 1, 3, 6, 9 and 12 month intervals in patients who were provided with a weaning schedule by the Neuromodulation team (experimental group) versus those who wean on their own or with their family doctor (control group; standard care) to determine if one strategy is superior to the other.

The secondary objectives will be to further characterize change in opioid use as it relates to pain scores, quality of life and disability from baseline to follow-up assessments. The investigators will examine changes in opioid-related adverse events and medication costs to help understand the impact of opioid weaning on the patient and the system. The investigators will also compare worker's compensation patients with non-worker compensation patients to see if they follow the same result pattern.

The main hypothesis is that administration of a patient- specific opioid weaning schedule by a pain-specific pharmacist will produce a greater reduction in opioid use in SCS patients post-implant compared to self-management/ family physician-assisted weaning schedule.

Study Design Population & Setting The study has a prospective, randomized, partial-crossover design. The estimated study recruitment duration will be a total of 2.5 years. Individual patient follow up will continue for 12 months post SCS-implant, for a total duration of 3.5 years.The study will take place in one site at the Regina General Hospital in Regina, SK. The study will initially enroll 150 patients who have been approved for and consented for SCS, currently taking opioid medications for pain control, who are willing to undergo opioid weaning. They also must be willing to be randomized to the Neuromodulation clinic weaning schedule group or the Self/Family Physician managed weaning group. The Self/Family Physician managed weaning group will experience standard care for the duration of the study. At the 6-month follow-up, participants in the control group will be allowed to cross over to the experimental group.

Patient Screening:

Patients will be screened for eligibility once they have been consented for an SCS procedure. Screening will be done by the study coordinators (Neuromodulation clinic staff) during a regular scheduled appointment at the clinic.

Once participants have met the inclusion/exclusion criteria for the study, they will be approached by the study coordinator for informed consent. Once consent is provided, all participants will be asked to complete the baseline assessment of medication use, pain, quality of life, disability and sleep patterns. (see section 6.0). A letter will be sent to the patient's family physician informing him/her that their patient is participating in the study. If they are in the experimental group, the physician will be informed that the patient will be following an opioid weaning schedule developed and followed up by the Neuromodulation clinic. For the control group, the physician will be informed about the study, but the hypothesis and patient allocation group will be concealed so as not to bias standard of care for weaning in the control group.

Randomization After consent is obtained and prior to SCS implantation, participants will be randomly assigned to the experimental or control group using a computerized random number generator to allocate patients in a 1:1 ratio to the experimental group (Neuromodulation clinic weaning schedule) or control group (Self/Family physician weaning schedule). The randomization sequence table will be generated by a biostatistician in the Regina Qu'Appelle Health Region (RQHR). The group allocation for each patient will be sent to the study coordinator in sealed, opaque sequentially numbered envelopes to be opened after patients have been enrolled in the study. At this time, it is not feasible to randomly assign patients to a self-management weaning or to their family physician, therefore the investigators are comparing the experimental group to standard care. If possible, the investigators will perform a subgroup analysis to see if there are any differences between the self-management or family physician weaning individuals.

Blinding The surgeon and Neuromodulation clinic pharmacist will be blind to allocation of patients to the experimental or control group. Any updates to the schedule that are required for patients in the experimental group will be performed by the Neuromodulation clinic pharmacist. As part of current routine care, the pharmacist will sometimes modify patient's schedules. The patient won't be directly identified as a study participant. The patient will not be blinded as they will have direct interaction with their weaning schedule and physicians. The family physician for patients in the experimental group will not be blind, but will be asked to allow the Neuromodulation clinic to handle the opioid weaning. The physicians for the control group will not be told the patient's allocation but may guess the group so there will not be true blinding. Participants will be asked not to disclose their study group when interacting with the Neuromodulation clinic pharmacist. The statistician analyzing the data will be blinded to the group allocation until after the initial analyses are complete.

Neuromodulation Clinic Weaning Schedule & Amendments The Neuromodulation clinic pharmacist will develop a weaning schedule for all patients enrolled in the study to ensure there is no bias in the generation of the schedule for the experimental group. However, schedules will not be given to the control participants. Schedules will be individualized taking into account the amount of opioid, duration of opioid use, other adjunctive medications, and specific variables related to the patient. Amendments to the schedules will occur on follow up. Amendments will be written up and submitted to the Neuromodulation nurse who is not blinded. Only patients in the experimental group will have their amendments forwarded to both themselves and their physicians.

Sample size Approximately 50 patients per year are referred for either spinal cord or peripheral SCS implant in the RQHR. The investigators plan to approach all patients that meet the inclusion/exclusion criteria for a period of 2.5 years to enroll 150 patients with an expected attrition rate of 20% during the internalization period and 20% during the follow-up, leaving a final sample of 100 patients for analysis.Based on minimally clinically significant effects, to observe a reduction in number of opioid medications from baseline to 6-month follow-up, a sample size of 100 patients would be sufficient to detect a mean difference of 2 medications with a standard deviation of 5 with 80% power. To detect a 20% increase in the experimental group in the proportion of patients that reach a 30% reduction in opioid dose from baseline to 6 month follow-up compared to the control group, at least 93 participants would be needed with 80% power.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be taking at least 1 opioid for a minimum of 6 months
* Subject is a candidate for spinal cord stimulation procedure

Exclusion Criteria:

* Palliative
* Documented substance abuse
* Subject less than 18 years of age
* Subject is unwilling or unable to attend required visits and/or comply with study requirements
* Subjects are unable to undergo study assessments or complete questionnaires independently i.e.: illiterate
* Subject has enrolled or plans to enroll in any study that might confound the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Change in number of opioids from baseline to post-intervention at 6-months follow-up | baseline to 6 months followup

SECONDARY OUTCOMES:
Proportion of patients that reach a 30% reduction in opioid dose (morphine-equivalent) from baseline to post-intervention at 6-months follow-up | baseline to 6-months followup
Change in Number of opioids used at 1, 3, 9 and 12 months follow-up | baseline and 1, 3, 9 and 12 months followup
Change in Mean dose of opioids at 1, 3, 6, 9, 12 months follow up | baseline and 1, 3, 6, 9 and 12 months followup
Proportion of patients that reach a 30% reduction in opioid dose (morphine-equivalent) from baseline to post-intervention at 1, 3, 9 and 12 months follow-up | baseline and 1, 3, 9 and 12 months followup
Change in visual analogue pain (VAS) score | baseline and 1, 3, 6, 9 and 12 months followup
Change in Euroqol 5D (EQ-5D) score | baseline and 1, 3, 6, 9 and 12 months followup
Change in 36-item short form survey (SF-36) score | baseline and 1, 3, 6, 9 and 12 months followup
Change in Oswestry Disability Index (ODI) score | baseline and 1, 3, 6, 9 and 12 months followup
Change in Pittsburgh Sleep Quality Index (PSQI) score | baseline and 1, 3, 6, 9 and 12 months followup
Change in medication costs ($) | baseline and 1, 3, 6, 9 and 12 months followup
Number of opioid-related adverse events | baseline and 1, 3, 6, 9 and 12 months followup

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Buwembo, MD, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Regina General Hospital, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided